CLINICAL TRIAL: NCT05861557
Title: A Prospective Phase II Trial to Evaluate the Safety and Efficacy of Neoadjuvant Radiotherapy Combined With Immunotherapy for Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Neoadjuvant Radiotherapy Combined With Toripalimab for Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Zhou Huifang, Director of Otorhinolaryngology Department, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023HNRT01
Record Dates: First submitted 2023-04-27; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — toripalimab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Toripalimab + SBRT radiotherapy
  Interventions: Drug: Toripalimab; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Toripalimab — 240mg, Q3W，I.V., D1, 2 cycles (1cycle of toripalimab before and after the SBRT radiotherapy, respectively), followed by the maintenance of toripalimab for 6 months after the surgery.
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Subjects were treated with SBRT radiotherapy (8Gy*5Fx), after 1 cycle of immunotherapy

SUMMARY:
This is a phase II study. Twenty-three patients with locally advanced head and neck squamous cell carcinoma were planned to be enrolled to assess the efficacy and safety of neoadjuvant immunotherapy combined with radiotherapy.

DETAILED DESCRIPTION:
After receiving one cycle of immunotherapy, the subjects underwent SBRT radiotherapy to the lesion, followed by another cycle of immunotherapy. Surgery was performed 3-6 weeks later, and subsequent radiotherapy or chemoradiotherapy was decided after surgery based on pathological examination. Immunotherapy was maintained for 6 months. Treatment continued until disease progression, death, unacceptable toxicity, withdrawal of consent, or study termination by the principal investigator, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent;
* Age ≥ 18 years, regardless of gender;
* Histology or cytology confirmed head and neck squamous cell carcinoma, HNSCC (Oral cavity, oropharynx, larynx and hypopharynx), and previously untreated;
* Imaging confirmed that HNSCC was locally advanced and operable;
* Imaging confirmed no metastasis;
* ECOG physical status score 0-1;
* Life expectancy at least 24 weeks;
* Have measurable lesions;
* Good function of other major organs (liver, kidney, blood system, etc.):

Absolute neutrophil count ((ANC) ≥ 1.0×10^9), platelet (≥ 80×10^9), hemoglobin (≥ 80g/L). Blood biochemical examination must meet: serum creatinine (Cr) ≤1.5 times the upper limit of normal (ULN) or endogenous creatinine clearance ≥60mL/min; TBIL≤1.5×ULN; ALB≥30g/L; ALT and AST≤ 3.0×ULN; TSH≤1.5×ULN;

* Female patients with fertility must undergo a pregnancy test (serum or urine) within 14 days before enrollment, and the result is negative, and they voluntarily adopt appropriate methods of contraception during the observation period and within 120 days after the last administration; Male patients must voluntarily take effective contraceptive measures from the start of treatment until 120 days after the last administration.

Exclusion Criteria:

* Pregnant or breastfeeding, or planning to become pregnant during the study period
* Patients with active autoimmune diseases or immunodeficiency diseases, including but not limited to myasthenia gravis, interstitial pneumonia, enteritis, autoimmune hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, positive HIV test or a history of the above diseases, or a history of organ transplantation;
* Receiving systemic immunosuppressive drugs within 2 weeks before starting study treatment, or anticipating the need for systemic immunosuppressive drugs during study treatment;
* Received systemic immunostimulants (including but not limited to interferon or interleukin-2 [IL-2]) within 4 weeks before starting study treatment;
* History of other malignant tumors within the past 5 years, except cured cervical carcinoma in situ, non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ;
* Serious cardiovascular disease, unstable arrhythmia, or unstable angina pectoris within 3 months before starting study treatment;
* The subject has an active infection or infectious disease, or unexplained fever (body temperature > 38.5℃) during screening and before the first dose;
* Patients who have received therapeutic oral or intravenous antibiotics within 2 weeks prior to starting study treatment; patients receiving prophylactic antibiotic therapy (e.g., prophylaxis for urinary tract infection or chronic obstructive pulmonary - Untreated active hepatitis;
* Receiving immunotherapy such as PD-1/L1 antibody or CTLA-4 antibody within 4 weeks before enrollment;
* Received chemotherapy or targeted therapy within 4 weeks before enrollment;
* The subject has participated in or completed other clinical trials within 4 weeks before enrollment;
* Subjects may need to receive other anti-tumor therapy during the study;
* Subjects may need to receive a vaccine during the study or within 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) | up to 6 months
  Percentage of Participants with MPR. MPR is defined as > 90 percent decrease in viable tumor.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) | up to 6 months
  Percentage of Participants with pCR. pCR is defined as the absence of residual tumor in both primary tumor and lymph nodes after neoadjuvant treatment.
Frequency and severity of perioperative adverse events | up to 6 months
  Grade 2-5 AEs according to NCI-CTCAE V5.0
Quality of life questionnaires | up to 1 year
  EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Huifang Zhou, Principal Investigator — Tianjin Medical University General Hospital; Ximei Zhang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (2):
- China (2):
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin